CLINICAL TRIAL: NCT01573052
Title: Comparison of Chlordiazepoxide and Gabapentin for Outpatient Alcohol Detoxification Treatment
Brief Title: Gabapentin vs Chlordiazepoxide for Ambulatory Alcohol Withdrawal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: VA Salt Lake City Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Christopher J. Stock, PharmD, Investigational pharmacist, VA Salt Lake City Health Care System
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UU40574
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2020-08-17 (Actual); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Withdrawal
MeSH Terms: interventions — Chlordiazepoxide; Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlordiazepoxide (Active Comparator): Chlordiazepoxide 25mg capsule or matching placebo capsule
  Interventions: Drug: Chlordiazepoxide
- Gabapentin (Experimental): Gabapentin 300mg capsule or matching placebo capsule
  Interventions: Drug: Gabapentin

INTERVENTIONS:
Drug: Chlordiazepoxide — 25mg four times daily x 3 days then tapered over 3 days
  Other Names: Librium
  Arms: Chlordiazepoxide
Drug: Gabapentin — 300mg four times daily x 3 days then tapered over 3 days
  Other Names: Neurontin
  Arms: Gabapentin

SUMMARY:
A randomized, double-blind controlled trial comparing treatment outcomes between chlordiazepoxide, or gabapentin to treat alcohol withdrawal syndrome in alcohol dependent veteran subjects. The objective of this trial is to compare the safety and effectiveness of these two medications. Intervention is a fixed dose taper of chlordiazepoxide, or gabapentin over 6 days. Subjects will be evaluated for 7-10 days to monitor alcohol abstinence, withdrawal severity scores, adverse events including ataxia, sedation, cognitive function and alcohol craving.

DETAILED DESCRIPTION:
Chlordiazepoxide 25 mg and matching placebo capsules or gabapentin 300 mg and matching placebo capsules were were used. The chlordiazepoxide/placebo and gabapentin/placebo capsules were not identical in appearance. Study medications were packaged into a 7-day medication organizer. The dosing for each subject was either gabapentin 1200mg or chlordiazepoxide 100 mg orally days 1-3, gabapentin 900 mg or chlordiazepoxide 75 mg day 4, gabapentin 600 mg or chlordiazepoxide 50 mg day 5, and gabapentin 300 mg or chlordiazepoxide 25 mg day 6.

Adherence was assessed by pill counts and serum samples were obtained for study drug analysis. Serum samples were batched and sent to a contract laboratory so that study clinicians were blinded to the results until after the trial was completed. Presence of the assigned study medication in the blood served as a surrogate adherence marker.

Subjects also received prescriptions for daily oral therapeutic multiple vitamin tablets, folic acid 1 mg, and thiamine 100 mg.

A psychiatric history and physical examination, breath alcohol concentration, vital signs, CIWA-Ar (alcohol withdrawal scale), and blood chemistry including transaminases and complete blood cell count were obtained for baseline for all participants. Subjects were seen on weekdays for clinic follow-up appointments. Assessments performed at each study visit included CIWA-Ar, ESS (Epworth Sleepiness Scale), PACS (Penn Alcohol Craving Scale), and a brief examination to document mental status and assess coordination, which included assessment of stance, tandem gait, Romberg test, pronator drift, toe and heel walk, rapid-alternating-movements, and point-to-point movements. Breath alcohol concentration (BAC) was also measured (AlcoSensor, Intoximeters, Inc.) at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Alcohol dependent at risk for withdrawal symptoms

Exclusion Criteria:

* Benzodiazepine dependent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2004-03; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Stock, PharmD, Principal Investigator — Salt Lake VA Health Care System
Locations (1):
- George E Wahlen VA Medical Center, Salt Lake City, Utah, United States

REFERENCES:
- [Derived] Stock CJ, Carpenter L, Ying J, Greene T. Gabapentin versus chlordiazepoxide for outpatient alcohol detoxification treatment. Ann Pharmacother. 2013 Jul-Aug;47(7-8):961-9. doi: 10.1345/aph.1R751. Epub 2013 Jun 18. PMID 23780805

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from VA outpatient detoxification clinic
Pre-assignment Details: Exclusions: subjects requiring hospitalization, receiving benzodiazepines prior to randomization and subjects not likely to follow instructions.
Groups:
- Chlordiazepoxide: 25mg four times daily x 3 days, 25mg three times daily x 1 day, 25mg twice daily x 1 day, 25mg at bedtime x 1 day then discontinue
- Gabapentin: 300mg four times daily x 3 days, 300mg three times daily x 1 day, 300mg twice daily x 1 day, 300mg at bedtime x 1 day then discontinue
Period: Overall Study
Arm/Group | Chlordiazepoxide | Gabapentin
Started | 9 | 17
Completed | 6 | 11
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Chlordiazepoxide: 25mg qid x 3 days, 25mg tid x 1 day, 25mg bid x 1 day, 25mg hs x 1 day then d/c
- Gabapentin: 300mg qid x 3 days, 300mg tid x 1 day, 300mg bid x 1 day, 300mg hs x 1 day then d/c
- Total: Total of all reporting groups
Arm/Group | Chlordiazepoxide | Gabapentin | Total
Number analyzed (Participants) | 9 | 17 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.8 (4.8) | 51.1 (7.7) | 52.7 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 8 | 17 | 25

OUTCOME MEASURES:

1. Primary Outcome: Epworth Sleepiness Scale (ESS)
Description: ESS is an 8 item-scale and scores range between 0 and 24. The higher the score implies more daytime sleepiness.
Time Frame: 1 week
Population: Late withdrawal period days 5-7
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chlordiazepoxide | Gabapentin
Number analyzed (Participants) | 9 | 17
units on a scale | 6.35 [3.13 to 9.57] | 2.65 [0.44 to 4.85]

2. Primary Outcome: PENN Alcohol Craving Scale
Description: PENN is a 5 item self-rated scale of alcohol craving. Scores range from 0 (little craving for alcohol) to 30 (irresistable urge to drink alcohol)
Time Frame: 1 week
Population: Late withdrawal period days 5-7
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Chlordiazepoxide | Gabapentin
Number analyzed (Participants) | 9 | 17
units on a scale | 16.78 [10.92 to 22.64] | 10.74 [7.09 to 14.39]

3. Secondary Outcome: Clinical Institute Withdrawal Assessment-Alcohol (Revised)(CIWA-Ar)
Description: CIWA-Ar measures severity of 10 observed or measured alcohol withdrawal signs or symptoms. Total score ranges from 0 (best possible outcome)-67 (worst possible outcome). Many previously publications suggest a total score of 8-10 is severe enough to warrant medication treatment. Lower scores (0-8) represent fewer withdrawal symptoms and less severity, scores > 8 represent more withdrawal symptoms and greater severity
Time Frame: 1 week
Population: Late withdrawal period days 5-7
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Gabapentin: 300mg four times a day x 3 days, 300mg three times daily x 1 day, 300mg twice daily x 1 day, 300mg at bedtime x 1 day then discontinue
Arm/Group | Chlordiazepoxide | Gabapentin
Number analyzed (Participants) | 9 | 17
units on a scale | 3.29 [-0.28 to 6.88] | 4.33 [2.10 to 6.56]

ADVERSE EVENTS:
Time Frame: 7 days
Description: Daily assessments of mental status, stance, tandem gait, Romberg test, pronator drift, toe and heel walk, rapid-alternating-movements, and point-to-point movements.
Arm/Group | Chlordiazepoxide | Gabapentin
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/17
Other Adverse Events (participants affected / at risk) | 0/9 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No